CLINICAL TRIAL: NCT05443529
Title: L'activitié Physique Sportive organisée Pour Sujets en Situation de Handicap : Impact Chez Les Sujets Post-accident Vasculaire cérébrale, Sur Les Trois Domaines de la Classification Internationale du Fonctionnement, du Handicap et de la santé (CIF)
Brief Title: Adaptive Sports for Individuals With a Physical Disability : Effect Among Stroke Survivors
Acronym: APSA-AVC
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Cliniques universitaires Saint-Luc- Université Catholique de Louvain (Other)
Responsible Party: Sponsor
Other Study IDs: 2022/13AVR/164
Record Dates: First submitted 2022-06-23; First posted 2022-07-05 (Actual); Last update posted 2023-11-24 (Actual); Status verified 2023-11

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Adaptive sports group: Individuals with stroke who regularly, and on a long-term basis, participate in adaptive sports
  Interventions: Other: Adaptive sports
- Non adaptive sports group: Individuals with stroke who do not engage in adaptive sports

INTERVENTIONS:
Other: Adaptive sports — Participation in community adaptive sports programs
  Groups: Adaptive sports group

SUMMARY:
The objective of the study is to evaluate the effect of engaging in adaptive sports for individuals who have had a stroke. The study is cross-sectional, participants with stroke will be recruited and divided into two groups: the first group composed of individuals with stroke who regularly participate in adaptive sports; and the second of individuals with stroke who do not regularly participate in adaptive sports. The two groups will have to be similar in terms of demographic variables (age, gender, time since beginning of stroke). A series of parameters will be tested, on one occasion for each participant. The two groups will then be compared to one another.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of stroke since at least 6 months prior to recruitment in the study
* persistent physical disability due to the stroke
* adequate understanding of french

Exclusion Criteria:

* significant cognitive impairments
* contra-indication of any type to performing physical activity and physical exercise

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population are individuals with a stroke diagnosis since a minimum of 6 months prior to the study. These individuals have to present persistent physical disability due to their stroke. The investigators will recruit individuals with stroke who participate in organised adaptive sports programs on a regular basis, as well as individuals who do not participate in any oranised adaptive sports programs.
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2022-10-18 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Functional walking | baseline
  Measured through a 6 minute-walk test where participants walk back and forth from one cone to another (placed 30 meters away), during 6 minutes. The distance walked in the 6 minutes is calculated.

SECONDARY OUTCOMES:
Physical endurance | baseline
  Measured through a sub-maximal effort test on cycle ergometer.
Motor impairment | baseline
  Measured by the Fugl-Meyer Assessment. The score ranges from 0-226, where lower scores represent greater motor impairment.
Upper and lower limb strength | baseline
  Measured using a manual dynamometer (microfet), in flexion, extension, adduction, abduction, internal rotation and external rotation of each limb.
Functional autonomy | baseline
  Measured using the Functional Independence Measure. Total scores range from 8 to 126 points. A lower score corresponds to complete dependence/no autonomy.
Functional walking capacity | baseline
  Measured by the timed up and go test.
Functional walking speed | baseline
  Measured by the 10 meter walk test.
Locomotion ability | baseline
  Measured by the Abiloco questionnaire. Score ranges from 0 to 13, where lower scores represent loss locomotion ability.
Balance | baseline
  Measured by the Activities-specific balance confidence scale. Scores range from 0 to 160, where higher score mean better confidence in balance.
Physical activity level (subjective) | baseline
  Measured by the Physical activity scale for individuals with physical disabilities. Scores range from 0 to 199.5 MET hour per day, where a greater score represents a greater level of physical activity.
Volume of physical activity performed daily | baseline, during one week
  Measured by an accelerometer.
Fatigue | baseline
  Measured by the fatigue severity scale. Scores range from 9 to 63 where a higher score represents greater fatigue severity.
Satisfaction with quality of life | baseline
  Measured by the EUROHIS-QOL (European Health Interview Survey, Quality of Life) 8 item questionnaire. Scores range from 0 to 40, with a greater score representing a better quality of life.
Social participation | baseline
  Measured by the Return to normal living index, a scale ranging from 0 to 100, with a greater score for greater social participation.
Intensity of physical activity performed daily | baseline, during one week
  Measured by a heart rate monitor

OTHER OUTCOMES:
Demographic variables | baseline
  Questionnaire asking participants to report age, gender, date of stroke, type of stroke as well as number of weekly sessions in any type of organised physical activity.
Medical and paramedical data | baseline
  Questionnaire asking participants to report any medication taken at the time of study participation, number of weekly sessions of physiotherapy and number of weekly sessions of other therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Gaëtan Stoquart, MD, Principal Investigator — Cliniques universitaires Saint-Luc- Université Catholique de Louvain
Locations (1):
- Cliniques Universitaires Saint-Luc, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: Undecided